CLINICAL TRIAL: NCT07180316
Title: Comparison of the Occurrence of Postoperative Complications Between Robotic and Laparoscopic Surgery in Revision Bariatric Surgery
Acronym: ROLAP
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-06-033-ERAME0598
Record Dates: First submitted 2025-06-24; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Obesity and Overweight; Bariatric Surgery
Keywords: bariatric revision surgery.; Laparoscopy; Robotic surgery
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LAPAROSCOPY SURGERY
- ROBOTIC SURGERY

SUMMARY:
In a population of patients undergoing bariatric revision surgery with conversion to RYGB and divided into two groups according to the surgical protocol:

Group 1: robotic surgery Group 2: laparoscopy

The primary objective of the study is to compare the rates of postoperative complications between the two groups, classified according to the Clavien Dindo classification. The secondary objectives are to compare between the groups:

* Total duration of the surgical procedure, stay in the emergency room, and hospitalization
* Postoperative pain
* Adverse events
* Weight loss
* Improvement in comorbidities

DETAILED DESCRIPTION:
The study procedures are the usual procedures of investigators who usually perform bariatric revision surgery. There is no change from the usual care. Participation in the study does not alter the benefit/risk ratio of the surgical procedure, does not alter the usual follow-up of patients who have undergone this type of surgery, and does not collect data other than those usually collected as part of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years,
* Patients who have been informed of the objectives and conditions of the study and who have not objected to the collection of their data
* Patients who are candidates for or have undergone revision bariatric surgery with conversion to RYGB (post-ring, post-sleeve, post-OAGB)

Exclusion Criteria:

* Pregnant patient
* Patient unable to understand information: dementia, psychosis, impaired consciousness, language difficulties

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing revision bariatric surgery with conversion to RYGB
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication rate | 12 month
  The complications routinely screened for are: gastrointestinal fistulas (gastrojejunal anastomosis fistula, excluded gastric fistula, and loop foot fistula), bruit, anastomotic stenosis, anastomotic ulcer, splenic infarction, the development of a deep abdominal collection, and pulmonary and cardioembolic complications.
  The diagnosis of gastrointestinal fistula will be made in the event of signs of sepsis associated with the presence of an intra-abdominal collection on CT scan, the need for intravenous antibiotics with strict fasting and exclusive parenteral nutrition, and/or the need for surgical exploration.
  Depression is defined as the postoperative need for blood transfusion, with a drop in hemoglobin levels of at least 2.5 g/dL compared to the preoperative level. Postoperative complications will be obtained according to the Clavien Dindo classification

SECONDARY OUTCOMES:
Post-operative PAIN | Day 2
  Post-operative pain will be assessed by a simple numerical scale rated from 0 (no pain) to 10 (worst pain ever experienced).
The total duration of the surgical procedure | Day 2
  Duration of anesthesia, duration of the surgical procedure,Length of stay in the Post-Anesthesia Care Unit, Time from end of surgery to first mobilization, Time from end of surgery to hospital discharge will be collected and compared between the two groups.
Weight loss | 12 month
  BMI will be collected during follow-up, and weight loss will be compared between the two groups.
Evolution of comorbidities | 12 month
  The occurrence, worsening, or resolution of the following comorbidities will be recorded:
  * Diabetes: type 1 or type 2
  * Arterial hypertension
  * Dyslipidemia
  * Obstructive sleep apnea syndrome (OSAS) or other severe obesity-related respiratory disorders
  * Chronic osteoarticular conditions
  * NASH (non-alcoholic steatohepatitis) or other metabolic liver diseases
  * Metabolic syndrome (defined as the presence of at least three of the following metabolic abnormalities: increased waist circumference, hyperglycemia, hypertension, hypertriglyceridemia, low HDL cholesterol)
  * Nephropathy
  * PCOS (Polycystic Ovary Syndrome)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital privé de la Loire - Ramsay Santé, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No